CLINICAL TRIAL: NCT04632758
Title: An Open-label, Randomized, Multicenter Phase 3 Study Comparing WX-0593 to Crizotinib in Anaplastic Lymphoma Kinase (ALK) Positive Non-Small Cell Lung Cancer (NSCLC) Patients
Brief Title: Study Comparing WX-0593 to Crizotinib in ALK Positive Non-Small Cell Lung Cancer (NSCLC) Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WX0593-004
Record Dates: First submitted 2020-09-05; First posted 2020-11-17 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WX-0593 Tablets (Experimental): Eligible patients with ALK+ NSCLC will receive WX-0593 tablets without food until documented disease progression or unacceptable toxicity. 60 mg of WX-0593 tablets, once daily for 7 days, followed by 180 mg of WX-0593 tablets, once daily in a 28-days cycle.
  Interventions: Drug: WX-0593 Tablets
- crizotinib (Active Comparator): Eligible patients with ALK+ NSCLC will receive oral crizotinib at 250mg BID without food until documented disease progression or unacceptable toxicity.
  Interventions: Drug: crizotinib

INTERVENTIONS:
Drug: WX-0593 Tablets — tablets, 60 mg→180mg, QD
  Other Names: FL-006
  Arms: WX-0593 Tablets
Drug: crizotinib — Capsules, 250mg, BID
  Arms: crizotinib

SUMMARY:
The primary purpose of this study is to evaluate the efficacy and safety of WX-0593 vs. crizotinib in patients with ALK-positive non-small cell lung cancer who had not received prior systemic therapy

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of WX-0593 vs. crizotinib in patients with ALK-positive NSCLC who had not received prior systemic therapy, to obtain additional pharmacokinetic (PK) data from sparse PK sampling, to compare the quality of life (QoL) in patients receiving WX-0593 vs. crizotinib, to evaluate the status of exploratory biomarkers and correlate with clinical outcome, and to obtain germline DNA samples for possible pharmacogenetic analysis in the event that outliers with respect to efficacy, tolerability/safety, or exposure are identified.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years
2. Female or male
3. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
4. Life expectancy of at least 12 weeks.
5. At least one measurable lesion (according to RECIST v1.1)
6. Histologically or cytologically confirmed diagnosis of advanced or recurrent or metastatic NSCLC that is ALK-positive by an Abbott FISH assay in the central lab. Randomization will occur after ALK positive confirmation is received from the central lab or local test using an method including Abbott FISH、RT-PCR or Ventana IHC.
7. No brain metastasis, or asymptomatic brain metastasis, or symptomatic brain metastasis but stable for more than 4 weeks after treatment, and have stopped systemic hormone treatment (prednisone of > 10 mg/day or equivalent hormone) for more than 2 weeks
8. Patients must have normal function as defined: ANC≥1.5*10^9/L; PLT≥90*10^9/L, Hb≥90 g/L, Total Bilirubin （TBIL）≤1.5*Upper Limit of Normal（ULN） ( Gilbert's Syndrome TBIL ≤3.0*ULN and DBIL≤1.5*ULN )，Alanine Transaminase （ALT）and Aspartate Aminotransferase（AST）≤2.5*ULN. For liver metastasis patients, ALT and AST≤5*ULN, Cr≤1.5*ULN, LVEF≥50%.
9. Any surgery or prior radiation (expect for palliative radiation) /operations must have been completed at least 4 weeks prior to first dosing. Palliative radiation must have been completed at least 48 hours prior to first dosing.
10. Patients must be able to understand and volunteer to sign the informed consent.

Exclusion Criteria:

1. Patients that have previously received cancer therapy (i.e., other targeted therapies, chemotherapy, immunotherapy, biologic therapy, hormonal therapy).
2. Patients with tumor meningeal metastasis
3. Clinically significant cardiovascular disease within 6 months prior to first dosing.
4. Two consecutive corrected QT interval (QTc) > 480 ms through ECG examination during screening, ≥2 arrhythmias, ≥2 heart failure (according to CTCAE 4.03), atrial fibrillation and ventricular fibrillation of any grade, or clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention
5. Patients need medications that may prolong QT interval or induce torsades de pointes within 14 days prior to the first dosing or during the study.
6. Continuous use of corticosteroids for more than 30 days, or require chronic use of corticosteroids or other immunosuppressants
7. Past history of a large area of diffuse/interstitial pulmonary fibrosis, or known history of Grade 3 or 4 interstitial pulmonary fibrosis or interstitial lung disease.
8. Patients with Grade > 1 nausea, vomiting, or diarrhea (CTCAE 4.03), other GI dysfunction or GI disease that may potentially affect drug absorption.
9. Patients at risk for GI perforation or intestinal obstruction
10. Patient has received other investigational drug within 1 month prior to first dosing. Subject received other clinical trial treatment within 1 month prior to the first dose of the investigational drug.
11. Patients who are HBsAg-positive and/or HBcAB positive and HBV DNA > 103copies/mL, or HCV antibody-positive, or syphilis antibody- positive or known HIV infected.
12. Patients who cannot suspend the use of a strong CYP3A4 inducer or inhibitor at least 1 weeks prior to this study and during the study.
13. Patients who cannot suspend the use of a CYP3A4 substrate at least 1 weeks prior to this study and during the study, and the therapeutic index is low.
14. Females who are pregnant or breastfeeding. Pregnant or lactating female patients or a positive pregnancy test at baseline for females of childbearing potential.
15. Female patients who are unwilling to use effective contraceptive measures during the entire course of the study and within 6 months after the end of the study, or male patients who plan to have children.
16. Concurrent diseases that may seriously affect patient safety or impact patient completion of the study as determined by the investigator (such as clinically uncontrolled hypertension (blood pressure > 160/110 mmHg), severe diabetes, or thyroid disease).
17. Drug abusers and alcoholics. Drug or alcohol abuse. Alcohol abuse refers to drinking 14 units of alcohol per week: 1 unit = 285mL of beer, or 25mL of spirits, or 100mL of wine;
18. History of definitive neurological or mental disorder, including epilepsy or dementia
19. Patients with other malignant tumors within 5 years prior to screening (except for cured basal cell carcinoma of the skin, cervical carcinoma in situ, thyroid carcinoma in situ, and papillary thyroid carcinoma).
20. Patients with added risks associated with the study or may interfere with the interpretation of study results as determined by the investigator, or deemed unsuitable by the investigator and/or sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | from randomization until firstly recorded disease progression or death (whichever occurs earlier), or to the date that the last patients observed for 12 months
  PFS as assessed by independent radiology review based on RECIST v. 1.1 criteria

SECONDARY OUTCOMES:
Progression-free survival (PFS) | from randomization until firstly recorded disease progression or death (whichever occurs earlier), or to the date that the last patients observed for 12 months
  PFS based on investigator assessment
OS | from randomization until death due to any cause, withdraws informed consent, is lost to follow-up or refuses phone visits, or study completion（up to 2.5 years）
  Overall survival (OS)
Confirmed Objective Response Rate (ORR) Assessed By independent radiology review | From fist administration to the date that the last patients observed for 12 months
  ORR is defined the percentage of the participants who have achieved complete response (CR) or partial response (PR) per independent radiology review using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 after the initiation of study treatment.
Confirmed Objective Response Rate (ORR) Assessed By Investigators | From fist administration to the date that the last patients observed for 12 months
  ORR is defined the percentage of the participants who have achieved complete response (CR) or partial response (PR) per Investigators using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 after the initiation of study treatment.
Time to Response (TTR) Assessed By independent radiology | From fist administration to the date that the last patients observed for 12 months
  Assessed from date of the first dose until the date of progression per independent radiology review
Time to Response (TTR) Assessed By Investigators | From fist administration to the date that the last patients observed for 12 months
  Assessed from date of the first dose until the date of progression per investigator.
Duration of response (DOR) Assessed By independent radiology | From fist administration to the date that the last patients observed for 12 months
  The DOR is defined as the time from the date of the first response CR/PR (whichever is first recorded) to the date on which progressive disease (PD) is first noted or date of death.
Duration of response (DOR) Assessed By Investigators | From fist administration to the date that the last patients observed for 12 months
  The DOR is defined as the time from the date of the first response CR/PR (whichever is first recorded) to the date on which progressive disease (PD) is first noted or date of death.
CNS response rate based on independent radiology review | From fist administration to the date that the last patients observed for 12 months
  CNS response rate based on independent radiology review
CNS response rate based on investigator assessment | From fist administration to the date that the last patients observed for 12 months
  CNS response rate based on investigator assessment
Time to CNS progression | From fist administration to the date that the last patients observed for 12 months
  Time to CNS progression
Percentage of patients with adverse events | from the signing of the informed consent form until at least 28 days after the last dose of study drug was administered.
  the incidence of adverse events, including adverse events (AEs), serious adverse events (SAEs), treatment-emergent adverse events (TEAEs). Causality is determined by the investigator.
Plasma concentrations (Cssmin) | Cssmin before dosing on Cycle 1 Day 1, Cycle 1 Day 7, Cycle 1 Day 21, Cycle 2 Day 21, and Cycle 4 Day 21
  Minimum value of steady plasma-drug concentration for WX-0593 at participating sites
Patient reported time to deterioration (TTD) | From fist administration to the date that the last patients observed for 12 months
  Patient reported time to deterioration (TTD) as measured by EORTC C30/LC13 QoL questionnaire
Patient reported time to deterioration (TTD) | From fist administration to the date that the last patients observed for 12 months
  Patient reported time to deterioration (TTD) as measured by Lung Cancer Symptom Scale (LCSS) questionnaire
Patient reported health-related quality of life (HRQoL) | From fist administration to the date that the last patients observed for 12 months
  Patient reported health-related quality of life (HRQoL) as measured by EORTC C30/LC13 QoL questionnaire
Patient reported health-related quality of life (HRQoL) | From fist administration to the date that the last patients observed for 12 months
  Patient reported health-related quality of life (HRQoL) as measured by Lung Cancer Symptom Scale (LCSS) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Shi Y, Chen J, Yang R, Wu H, Wang Z, Yang W, Cui J, Zhang Y, Liu C, Cheng Y, Liu Y, Shan J, Wang D, Yang L, Hu C, Zhao J, Cao R, Tan B, Xu K, Si M, Li H, Mao R, Li L, Kang X, Wang L. Iruplinalkib (WX-0593) Versus Crizotinib in ALK TKI-Naive Locally Advanced or Metastatic ALK-Positive NSCLC: Interim Analysis of a Randomized, Open-Label, Phase 3 Study (INSPIRE). J Thorac Oncol. 2024 Jun;19(6):912-927. doi: 10.1016/j.jtho.2024.01.013. Epub 2024 Jan 25. PMID 38280448